CLINICAL TRIAL: NCT00086541
Title: A Phase 3, Randomized, Open-Label Study of the Safety and Efficacy of Two Dose Levels of Interferon Alfacon-1 (Infergen, CIFN) Plus Ribavirin Administered Daily for 48 Weeks Versus No Treatment in Hepatitis C Infected Patients Who Are Nonresponders to Previous Pegylated Interferon Alfa Plus Ribavirin Therapy
Brief Title: Daily-Dose Consensus Interferon and Ribavirin: Efficacy of Combined Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRHC-001; DIRECT 1
Record Dates: First submitted 2004-07-02; First posted 2004-07-07 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Liver; Pegylated; Interferon; Alpha; Ribavirin; Combination; Nonresponder; HCV; Infergen; SVR
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — interferon alfacon-1; Ribavirin

INTERVENTIONS:
Drug: Daily Infergen (Interferon Alfacon-1, CIFN) (9 or 15 µg) + Ribavirin (1000-1200 mg, based on body weight) PO Daily for up to 48 wks

SUMMARY:
This Phase 3 clinical study is designed to evaluate the safety, tolerability, and efficacy of two dose levels of Infergen (interferon alfacon-1, CIFN) plus Ribavirin administered daily for 48 weeks and no treatment in patients chronically infected with hepatitis C who are nonresponders to previous pegylated interferon alfa plus ribavirin therapy.

Patients are randomized 1:1:1 to receive Interferon Alfacon-1 (9 or 15 µg) + Ribavirin (both administered daily) or no treatment for up to 48 weeks.

The protocol and informed consent form that will be used must be approved by the Investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC) before the study is initiated.

ELIGIBILITY:
(Abbreviated due to space constraints.)

Inclusion Criteria:

1. Signed informed consent form
2. Male or female 18 yrs. of age or older
3. Chronic HCV infection based on documented history of positive serum anti-HCV antibody test and/or detectable levels of HCV RNA
4. Documented virologic nonresponse to past treatment with PEGASYS plus ribavirin or PEG-Intron plus ribavirin
5. Previously treated w/either of the following starting doses of pegylated interferon alpha:

   1. ≥ 1.5 µg/kg/week PEG-Intron or dose consistent with the package insert or,
   2. ≥ 180 µg/week PEGASYS
6. Detectable plasma HCV RNA level at screening visit
7. Liver biopsy histologically documenting chronic liver disease consistent with chronic HCV infection
8. All patients and all potentially fertile sexual partners of patients must use 2 reliable forms of effective contraception during the study & for 6 months after cessation of the study drugs

Exclusion Criteria:

1. Any history of decompensated liver disease
2. Any of a variety of laboratory abnormalities assessed through blood sample at screening
3. Patients who prematurely discontinued, interrupted, or reduced the dose of their previous pegylated interferon alpha-based combination therapy due to noncompliance or safety and/or tolerability issues
4. Patients who had undetectable HCV RNA levels during prior pegylated interferon alfa plus ribavirin treatment but who relapsed during follow-up
5. Significant depression in the last 2 years
6. Patients treated for HCV infection within 3 months before screening (w/the exclusion of over-the-counter therapies)
7. Patients who have been on any experimental protocol or therapy within 28 days before screening
8. Use of colony-stimulating factor agents or other therapeutic agents that might artificially elevate laboratory parameters within 3 months before screening
9. Known human immunodeficiency virus (HIV) infection or positive HIV antibody test at screening
10. Chronic hepatitis B infection or positive hepatitis B surface antigen (HBsAg) at screening
11. New onset diabetes
12. Unstable or uncontrolled thyroid disease
13. Presence or history of non-HCV chronic liver disease
14. History of unstable or deteriorating cardiac or cerebrovascular disease within 6 months before Screening
15. Current or history of neurologic disorder within the last 2 years
16. History of seizures within the past 5 years
17. History of hemoglobinopathies
18. History of malignancy within the last 5 years with the exception of localized basal or squamous cell carcinoma & fully resected, localized malignancy not requiring active treatment & with no evidence of recurrence
19. A disease known to cause significant alteration in immunologic function including hematologic malignancy, sarcoidosis or autoimmune disorder
20. History or evidence of retinopathy
21. History of major organ transplantation with an existing functional graft
22. Concurrent therapy with immunosuppressive drugs or cytotoxic agents
23. Alcohol and/or drug abuse w/in the past year, that in the opinion of the Investigator or the Sponsor may negatively affect patient compliance
24. Pregnant or lactating women
25. Male partners of women who are pregnant
26. Known sensitivity to Infergen or IFN-α or to E. coli-derived products
27. Patients who, in the opinion of the Investigator or the Sponsor, are not suitable candidates for enrollment or who would not comply w/the requirements of the study
28. Patients who have not responded to a course of daily Infergen (9 or 15 µg) with or without ribavirin or who have relapsed after a course of daily Infergen (9 or 15 µg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2004-06; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Evaluate sustained virologic response (SVR) rate of daily Infergen at two dose levels plus ribavirin and no treatment in chronically HCV-infected patients who are nonresponders to previous pegylated interferon alfa plus ribavirin therapy.

SECONDARY OUTCOMES:
Evaluate safety & tolerability of therapy detailed in primary objective, and proportion of patients with (a) undetectable plasma HCV RNA levels at weeks 24 & 48 (b) abnormal baseline serum ALT levels that are normal at week 24, week 48 and weeks 48 & 72.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph T. Doyle, Study Director — Bausch Health Americas, Inc.

REFERENCES:
- See also: Daily-Dose Consensus Interferon and Ribavirin: Efficacy of Combined Therapy — http://www.directtrial.com